CLINICAL TRIAL: NCT00739713
Title: Effects of Sea Buckthorn Oil on Dry Eye
Acronym: DESB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Turku Municipal Health Department/evo-funding (Unknown); Turku University Hospital (Other Government); Finnsusp Ltd. (Industry); Aromtech Ltd. (Industry); Shiny Horse Ltd (Unknown); Valioravinto Ltd (Unknown); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Matti Viitanen/ Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DESB
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2017-03

CONDITIONS: Dry Eye Syndromes
Keywords: dry eye; sea buckthorn; Hippophaë
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB (Experimental): Sea buckthorn oil group
  Interventions: Dietary Supplement: Sea buckthorn (Hippophaë rhamnoides) oil
- PL (Placebo Comparator): Placebo group
  Interventions: Dietary Supplement: Placebo comparison

INTERVENTIONS:
Dietary Supplement: Sea buckthorn (Hippophaë rhamnoides) oil — Dosage 2 g/d, frequency twice/d, duration 3 months
  Arms: SB
Dietary Supplement: Placebo comparison — Placebo comparison, dosage 2 g/d, frequency twice/d, duration 3 months
  Arms: PL

SUMMARY:
The objective is to study the effect of sea buckthorn oil on dry eye.

DETAILED DESCRIPTION:
The objective is to study whether regular consumption of sea buckthorn berry oil can relieve the symptoms of dry eye syndrome. The study design is a parallel randomized double-blind placebo controlled trial. The participants daily consume sea buckthorn or placebo oil for 3 months. The dry eye symptoms will be monitored during the study using a validated questionnaire. In addition clinical dry eye tests are made by an ophthalmologist three time during the study. Samples will be taken for tear film lipid and cytokine analyses. Blood samples for the analyses of inflammatory markers are also obtained. The cytokine and other inflammation marker analyses are optional. The symptoms will be monitored and clinical tests made also 4 weeks after the participants have stopped consuming the study oils.

ELIGIBILITY:
Inclusion Criteria:

* Dry eye symptoms

Exclusion Criteria:

* Severe illness
* Anticholinergic drugs
* Smoking

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Symptom severity: symptom questionnaires and clinical dry eye tests | 3 months intervention + 1 month after the intervention

SECONDARY OUTCOMES:
Tear film lipid profile, tear cytokines, inflammation mediators in blood | 3 months intervention + 1 month after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Heikki P Kallio, Professor, Study Director — University of Turku
Locations (1):
- University of Turku, Turku, Finland

REFERENCES:
- [Background] Yang B, Kalimo KO, Mattila LM, Kallio SE, Katajisto JK, Peltola OJ, Kallio HP. Effects of dietary supplementation with sea buckthorn (Hippophae rhamnoides) seed and pulp oils on atopic dermatitis. J Nutr Biochem. 1999 Nov;10(11):622-30. doi: 10.1016/s0955-2863(99)00049-2. PMID 15539258
- [Result] Larmo PS, Jarvinen RL, Setala NL, Yang B, Viitanen MH, Engblom JR, Tahvonen RL, Kallio HP. Oral sea buckthorn oil attenuates tear film osmolarity and symptoms in individuals with dry eye. J Nutr. 2010 Aug;140(8):1462-8. doi: 10.3945/jn.109.118901. Epub 2010 Jun 16. PMID 20554904